CLINICAL TRIAL: NCT05479266
Title: Comparison of Muscle Energy Techniques and Myofascial Release on Low Back Pain Due to Sacroiliac Joint Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RIPHAH/FR&AHS/Letter-0976
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Sacroiliac Joint Dysfunction; Low Back Pain
Keywords: sacroiliac Joint Dysfunction; Muscle Energy Techniques; Myofascial Release; Pain; Disability; Range of Motion
MeSH Terms: conditions — Low Back Pain; Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle Energy Techniques (Experimental): Muscle Energy Techniques and Conventional Physical Therapy
  Interventions: Other: Muscle Energy Technique
- Myofascial Release (Experimental): Myofascial Release and Conventional Physical Therapy
  Interventions: Other: Myofascial release

INTERVENTIONS:
Other: Muscle Energy Technique — METS-Post isometric relaxation will be applied for piriformis, iliopsoas and hamstrings muscle. There will be three repetitions for each muscle, once per day and thrice a week for three weeks
  Other Names: Transcutaneous Electrical Nerve Stimulations and Hot pack
  Arms: Muscle Energy Techniques
Other: Myofascial release — Myofascial Release will be done for piriformis, iliopsoas and hamstrings muscle. There will be three repetitions for each muscle, once per day and thrice a week for three weeks
  Other Names: Transcutaneous Electrical Nerve Stimulations and Hot pack
  Arms: Myofascial Release

SUMMARY:
The aim of this research is to compare the effects of Muscle Energy Techniques and Myofascial Release on Lumbar Range of motion, pain and disability in patients of low back pain due to Sacroiliac Joint Dysfunction, Randomized controlled trials were done at a private clinic, The Health Professionals Bahria Town Phase 6, Islamabad. The Sample Size was 30. The subjects were divided into two groups, 15 subjects in Interventional group A receiving conventional physical therapy treatment alongside METs for hamstrings, iliopsoas and piriformis muscle while the other 15 subjects in Interventional group B receiving conventional physical therapy treatment with direct myofascial release of hamstrings, iliopsoas and piriformis muscle. study duration was of 6 months. Samling technique applied was non.probability sampling. Only females of age group 40-55 yrs having sacroiliac joint pain with limited lumbar range of motion were reduced. Tools used in the study were Numeric Pain Rating Scale(NPRS), Modified Oswestry Disability Index(MODI), Pelvic and bubble Inclinometer. Data was analyzed through SPSS 21.

DETAILED DESCRIPTION:
Sacroiliac joint is the most common source of low back pain affecting 70-85% of adults. Accordingly, 13-30% of patients with lower back pain have Sacroiliac joint dysfunction. The main mechanism for developing sacroiliac joint dysfunction includes different unidirectional pelvic shear force along with repetitive torsional force and inflammation which produces not only the lower back pain but also groin and gluteal pain. Muscle imbalances has also been sighted as possible cause of pain. This theory states that the sacroiliac joint itself is unaffected, but the musculature surrounding the sacroiliac joint is in form of dysfunction. This muscular imbalance could limit the flexibility of muscle of low back pain and ultimately begin a syndrome of chronic disuse culminating in decreased function and heightened pain. The use of a combination of tests showed a high sensitivity and specificity to indicate the presence of sacroiliac joint dysfunction that includes FABER, posterior shear and resisted abduction pain provocation tests.

Treatment of sacroiliac joint pain is variable and no set method or protocol of treatment has been found to be efficacious and reliable. Interventions to treat pain of SIJ dysfunction includes Non-steroidal Anti-Inflammatory drugs(NSAIDs), physical therapy, corticosteroid injections, osteopathic manipulations(manual medicine), radiofrequency denervation, sacroiliac joint belts and surgery. Muscle Energy Techniques is the most commonly used manual medicine techniques that depends on method of using low amplitude muscle contractions against resistance thinking that it would improve vascular circulation and have a positive influence on static and dynamic posture. this techniques was further modified by having patients use their muscles in a controlled position against a counterforce. Muscle energy techniques have several uses that can help increase muscle strength, increase range of motion(ROM) and decrease edema.

Myofascial release techniques(MFR) are another manual medicine technique that is described as 'designed to stretch and reflexively release patterned soft tissue( particularly the muscles and fascia) and joint related restrictions'. myofascial abnormalities may lead to connective tissue fibrosis, increased tissue stiffness and further movement impairment which may lead to low back pain chronicity.

In a study conducted by D. Sharma et al in 2014 on comparing the effects of muscle energy techniques and mobilizations in treating sacroiliac joint dysfunction focusing on piriformis, quadratus lumborum and erector spinae muscles, concluded that METs and mobilizations are both effective in treating chronic low back pain due to sacroiliac joint dysfunction. Outcomes were measured on first day and then after 1st and 2nd week from each subject, pain and disability by Visual Analogue Scale and Modified Oswestry Disability Index Questionnaire(MODI) In a randomized controlled trial conducted by Arguisuelas et al in 2017 for studying the effects of Myofascial release (MFR) for quadratus lumborum, psoas muscle, thoracolumbar fascia and lumbar paravertebral muscles in Non-specific chronic low back pain , it was concluded that myofascial release therapy produced a significant improvement in both pain and disability. Pain was measured by means of Short Form Mc Gill Pain Questionnaire (SF-MPQ) and Visual Analogue scale and disability measured with Roland Morris Questionnaire.

In another study conducted by Sabah et al in 2019 concluded that muscle energy techniques for iliopsoas, hamstrings, erector spinae and quadratus lumborum is an effective treatment for decreasing anterior pelvic tilting angle and reducing pain in patients with chronic SIJ dysfunction. The study findings revealed a statistical significant decrease of anterior pelvic tilting angle in group A(p<0.001), also a significant decrease in pain in the 2 groups compared with the pre-intervention values(p<0.001) In 2020, Faryal et al conducted a study in peshawar, concluded that muscle energy technique targeting quadratus lumborum, iliopsoas and piriformis muscle and maitland mobilizations are both effective in treating the chronic sacroiliac joint dysfunction in terms of decreasing pain and disability when using lumbopelvic stabilization exercises as an adjunct therapy with them.

In previous studies both muscle energy techniques and myofascial release therapy has been proven to be effective in treating chronic low back pain due to sacroiliac joint dysfunction. Currently to our knowledge there exists very weak evidence to which one technique can be proved to be more effective than the other. The purpose of this study is to compare the effects of both these therapies on pain and functional status in patients with sacroiliac joint dysfunction in addition to conventional physical therapy treatment protocols.

ELIGIBILITY:
Inclusion Criteria:Participants falling in this category would be recruited into the study.

* Subjects who have had sacroiliac joint pain and hypomobility for 3-6 months
* Muscle tightness
* Only Female Gender
* Age b/w 40-55 years
* Limited Lumber Range of motion (by Inclinometer) (normal ranges flexion: 60 degrees Extension: 35 degrees Side bending: 20 degrees)
* Pain more than 3 on Numeric pain rating scale only

Exclusion Criteria:

* history of systemic illness
* acute injury or fracture in the lower limbs
* any hip joint pathology/infection/malignancy
* previous hip surgery or recently received intra-articular injections
* spinal stenosis/spondylolisthesis/disc disease
* congenital spinal deformity
* hypermobility of sacroiliac joint

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 3rd week
  NPRS is an 11- point numeric scale with 0 representing one pain extreme (e.g no pain) amd 10 representing the other extreme (e.g worst pain imaginable), scores range from 1-10. the highest the score the greater the intensity of pain
Modified Oswestry Disability Index | 3rd week
  this questionnaire consists of 10 items addressing different aspects of function. Each itemis scored from 0-5, with higher values representing greater disability. The total score is multiplied by 2 and expressed as percentage. Fore each section the total possible score is 5.
Range of Motion(lumbar spine) | 3rd week
  Lumbar spine flexion, extension and sidebending will be measured with bubble inclinometer
pelvic tilting | 3rd week
  pelvic tilting will be measured with pelvic inclinometer

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Affan Iqbal, PhD, Principal Investigator — Riphah International University
Locations (1):
- The Health Professionals, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No